CLINICAL TRIAL: NCT02798198
Title: The Correlation Between the Pulmonary Function and Intrarenal Hemodynamics in 37 T2DM Patients in Early Period
Status: Completed | Type: Observational
Sponsor: Fourth People's Hospital of Shenyang (Other)
Responsible Party: Principal Investigator, Jin-song Kuang, Chief physician, Fourth People's Hospital of Shenyang
Other Study IDs: 20150908
Record Dates: First submitted 2016-05-30; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Diabetes group: 37 T2DM adults (diabetes group) without DKD
  Interventions: Other: T2DM
- Control group: 33 healthy adults (control group)
  Interventions: Other: T2DM

INTERVENTIONS:
Other: T2DM — T2DM without DKD

SUMMARY:
Objective: The main target of this study was to research the early changes in pulmonary function and intrarenal hemodynamics, then research the correlation between the pulmonary function and the renal hemodynamics in type 2 diabetes (T2DM) patients without diabetic kidney disease (DKD).

Method: 37 T2DM patients (diabetes group) without DKD and 33 healthy people (control group) were choosed to research early changes in pulmonary function and intrarenal hemodynamics, then research the correlation between the pulmonary function and the renal blood flow in T2DM patients, all having normal renal function. The primary endpoints were the pulmonary function parameters (VC%, FVC%, FEV1%, PEF%, MVV%, TLC%, FEV1/FVC%, DLCO%, and DLCO/VA%); the secondary endpoints were the intrarenal hemodynamic (bilateral kidney RI) in bilateral interlobular renal arteries were evaluated using; the tertiary endpoints were the biochemical variables: blood-fat (TC, HDL-C, LDL-C, and TG), renal function parameters (BUN, Cr, and GFR); in addition, the albumin excrete rate (AER), urinary albumin/creatinine ratio (UACR) were measured.

DETAILED DESCRIPTION:
Pulmonary function was measured by spirometer which was provided by Jaska Corporation in Japan, model number: HI-101; RI were measured by Logiq 400 MD Pro Series scanner (GE Medical Systems, Milwaukee, WI) using a 3.5-4 MHz vector array transducer

ELIGIBILITY:
Inclusion Criteria:

1) The patients were diagnosed with T2DM according to the guidelines of the American Diabetes Association ; 2) No smoking history, pulmonary disease, cold, nor pulmonary infection within a fortnight; 3) Did not have hepatopathy, nephropathy, hyperuricemia, and gastrointestinal disease; and 4) Likely to have good compliance and able to visit our hospital for periodic assessments.

Exclusion Criteria:

1) T1DM, gestation and lactation; 2) Renal inadequacy; 3) Hypohepatia; 4) Intensive care with insulin treatment; 5) The patients combinated with DKD and hypertension (antihypertensive drugs were used); 6) Patients with other renal conditions that could affect the hemodynamics, such as urolithiasis, urinary infection, and renal cyst (diameter > 3 cm); 7) Heart failure; 8) Cholesterol-lowering drugs can not control the blood-fat ; and 9) Use of systemically injected glucocorticoids within 3 months prior to our study.

Ages: 35 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We selected 42 T2DM patients (24 males, 18 females) without DKD as diabetes group and 38 healthy people (21 males, 17 females) as control group from the diabetic outpatient clinic in Shenyang the Fourth Hospital of People, but only 37 patients (21 males, 16 females) in the diabetes group and 33 healthy people (18 males, 15 females) can be researched in our study, all the participants were the Chinese Hans.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The pulmonary function (using spirometer) in the healthy people and T2DM patients and comparing the differences between the two groups | one week
  pulmonary function parameters include: VC%, FVC%, FEV1%, PEF%, MVV%, TLC%, FEV1/FVC%, DLCO%, and DLCO/VA%
The bilateral kidney RI(using CDI) in healthy people and T2DM patients and comparig the differences between the two groups | one week
  The Doppler resistance index (RI) [(peak systolic velocity, PSV - peak end diastolic velocity, PED)/ peak systolic velocity, PSV
The correlation between the pulmonary function and the renal hemodynamics in 37 T2DM patients without DKD | two weeks

SECONDARY OUTCOMES:
Blood-fat (TC, HDL-C, LDL-C, and TG)in the healthy people and T2DM patients and comparing the differences between the two groups | Three weeks
Renal function parameters (BUN, Cr) in the healthy people and T2DM patients and comparing the differences between the two groups | Three weeks
The albumin excrete rate (AER), urinary albumin/creatinine ratio (UACR)in the healthy people and T2DM patients and comparing the differences between the two groups | Three weeks

REFERENCES:
- [Derived] Tai H, Jiang XL, Kuang JS, Yu JJ, Ju YT, Cao WC, Chen W, Cui XY, Zhang LD, Fu X, Jia LQ, Zhang Y. Early changes in pulmonary function and intrarenal haemodynamics and the correlation between these sets of parameters in patients with T2DM. PLoS One. 2019 Dec 18;14(12):e0224923. doi: 10.1371/journal.pone.0224923. eCollection 2019. PMID 31851677